CLINICAL TRIAL: NCT02456376
Title: Sensor Fusion for Balance Control in Children With Cerebral Palsy
Brief Title: Balance Control in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Collaborators: Shriners Hospitals for Children (Other); University of Delaware (Other)
Responsible Party: Principal Investigator, John Jeka, Professor, Temple University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71002-PHI-14; 22173 (Other: Temple IRB)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Cerebral Palsy
Keywords: Sensor Fusion; Stochastic Resonance Stimulation; Sensory deficits; Postural Control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children with Cerebral palsy (Experimental): 1. Sensory integration testing
  2. SR stimulation and Sensory integration testing
  Interventions: Procedure: Sensory Integration Testing; Procedure: SR stimulation & Sensory integration testing
- Children with Typical Development (Active Comparator): 1. Sensory integration testing
  2. SR stimulation and Sensory integration testing
  Interventions: Procedure: Sensory Integration Testing; Procedure: SR stimulation & Sensory integration testing

INTERVENTIONS:
Procedure: Sensory Integration Testing — Investigate how sensory information are integrated during upright stance when visual and body senses are challenged in a virtual reality environment
  Other Names: Sensor Fusion paradigm
Procedure: SR stimulation & Sensory integration testing — Use SR stimulation to improve sensory integration when visual and body senses are challenged in a virtual reality environment

SUMMARY:
The purpose of this study is to investigate how sensory information processing affects balance ability in children with cerebral palsy (CP). An additional goal is to determine if a subsensory electrical stimulation called Stochastic Resonance (SR) Stimulation, can improve balance in children with CP. Children with CP and children with typical development will participate and complete a series of clinical and balance assessments. They will also be tested in a sensor fusion paradigm to investigate potential deficits in the dynamic integration of visual, vestibular and proprioceptive information during upright stance. SR stimulation will then be used to potentially improve these deficits and subsequently their balance ability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic diplegia CP (GMFCS I- III)*
* Ability to stand independently for approximately 2 min

Exclusion Criteria:

* Lower extremity surgery or fractures in the year prior testing
* Joint instability or dislocation in the lower extremities
* Botulinum toxin injections in the lower extremities within the past 6 months*
* Marked visual or hearing deficits
* Uncontrolled seizure disorder
* Implanted medical device that may be contraindicated with application of SR stimulation

  * Asterisk indicates the eligibility criteria that should be met only by children with CP

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Gain response | 1 day
  For both the sensory reweighting testing, the visual signal will be displayed as a visual flow with translation in anterior-posterior (AP) direction (i.e., sagittal plane) and presented at different amplitudes (0.25 and 0.5 cm) at 0.2 Hz to measure: the change in gain (weighting) to vision (intramodal effect); and a change in gain to vibration and galvanic stimulation (intermodal effects). Gain for each modality relative to both the leg segment AP translation and trunk segment AP translation will be measured.

SECONDARY OUTCOMES:
Gain response | 1 day
  For the sensory reweighting with the addition of SR stimulation testing, the visual signal will be displayed as a visual flow with translation in anterior-posterior (AP) direction (i.e., sagittal plane) and presented at different amplitudes (0.25 and 0.5 cm) at 0.2 Hz to measure: the change in gain (weighting) to vision (intramodal effect); and a change in gain to vibration and galvanic stimulation (intermodal effects). Gain for each modality relative to both the leg segment AP translation and trunk segment AP translation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: John Jeka, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Temple University, Philadelphia, Pennsylvania
  - Shriners Hospital for Children, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Zarkou A, Lee SCK, Prosser LA, Hwang S, Jeka J. Stochastic resonance stimulation improves balance in children with cerebral palsy: a case control study. J Neuroeng Rehabil. 2018 Dec 10;15(1):115. doi: 10.1186/s12984-018-0467-7. PMID 30526617